CLINICAL TRIAL: NCT02086162
Title: RCT of a Motivational Decision Support System for Smokers With Severe Mental Illnesses
Brief Title: Randomized Controlled Trial (RCT) of a Motivational Decision Support System
Acronym: RCTEDSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary F. Brunette, MD, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FED14095; R01CA168778 (NIH)
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Smoking; Tobacco; Motivation; Cessation Treatment
MeSH Terms: conditions — Schizophrenia; Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral intervention (Experimental): Web-based motivational decision support system
  Interventions: Behavioral: Web-based motivational decision support system
- Educational intervention (Active Comparator): Computerized version of the National Cancer Institute (NCI) Educational Pamphlet
  Interventions: Behavioral: NCI Education

INTERVENTIONS:
Behavioral: Web-based motivational decision support system
  Arms: Behavioral intervention
Behavioral: NCI Education
  Arms: Educational intervention

SUMMARY:
In this study we will definitively test the decision support system in a randomized controlled trial (RCT) among smokers with severe mental illness (SMI) psychotic disorders. The Specific Aims of the study are:

1. To determine whether use of the web-based decision support system leads to higher rates of initiation of smoking cessation treatment than use of a computerized educational pamphlet. We will also assess effectiveness on secondary outcomes, including smoking behavior, urges and outcome expectancies; level of dependence; intentions to quit and to use cessation treatment; and abstinence.
2. To assess whether cognitive ability moderates initiation of smoking cessation treatment. Since cognitive impairment impedes use of standard web-based interventions by this group, and cognitive impairments likely supersede other potential moderators (education and socioeconomic status), this aim will be key to determining the success of our intervention and will guide further revisions if they are needed.
3. To explore the effects of the decision support system and baseline cognitive ability on abstinence over 6 months

   1. We will examine the impact of the DSS on 7-day point prevalence tobacco abstinence at 6 months, and cumulative days of tobacco abstinence over 6 months.
   2. We will determine whether baseline cognition (scale scores) is associated with 7-day point prevalence tobacco abstinence at 6 months, and cumulative days of tobacco abstinence over 6 months.

DETAILED DESCRIPTION:
Up to 80% of people with schizophrenia and schizoaffective disorders smoke - a rate that is four times the rate in the general population. Cessation treatments are effective, but these smokers don't use them. In order to provide an easy-to-use, cost-effective strategy to engage this group of smokers into effective treatments, we developed a single-session, web-based, motivational decision support system, Let's Talk About Smoking. The system incorporates features that insure high usability among those who can't use current websites due to cognitive impairments and low computer skills. It provides compelling content that engages users into evidence-based cessation treatments.

In this study we will definitively test the decision support system in a randomized controlled trial (RCT) among smokers with severe mental illness (SMI) psychotic disorders. Our proposed study design will enable us to test whether this system, designed for those with cognitive impairments, is effective among people with a range of cognitive abilities. The Specific Aims of the study are:

1. To determine whether use of the web-based decision support system leads to higher rates of initiation of smoking cessation treatment than use of a computerized educational pamphlet. We will also assess effectiveness on secondary outcomes, including smoking behavior, urges and outcome expectancies; level of dependence; intentions to quit and to use cessation treatment; and abstinence.
2. To assess whether cognitive ability moderates initiation of smoking cessation treatment. Since cognitive impairment impedes use of standard web-based interventions by this group, and cognitive impairments likely supersede other potential moderators (education and socioeconomic status), this aim will be key to determining the success of our intervention and will guide further revisions if they are needed.
3. To explore the effects of the decision support system and baseline cognitive ability on abstinence over 6 months

   1. We will examine the impact of the DSS on 7-day point prevalence tobacco abstinence at 6 months, and cumulative days of tobacco abstinence over 6 months.
   2. We will determine whether baseline cognition (scale scores) is associated with 7-day point prevalence tobacco abstinence at 6 months, and cumulative days of tobacco abstinence over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* DSM-IV-TR diagnosis psychotic disorder
* in treatment at participating mental health center
* current daily smoker
* fluent in English
* physically able to use computer
* willing and able to give informed consent

Exclusion Criteria:

* past 2 weeks use of evidence based cessation treatment
* psychiatric instability
* current alcohol or drug dependence
* pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F. Burnette, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (3):
- United States (3):
  - Thresholds, Chicago, Illinois
  - University of Massachusetts, Worcester, Massachusetts
  - Rutgers-UNDMJ, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
De-identified research data files will be made available to all researchers in both the public and private sectors for potential statistical analyses or re-analyses in accordance with the NIH data Sharing Policy: http://grants.nih.gov/grants/policy/data sharing. Data will be available 2 years after data collection is completed, or after primary papers have been accepted for publication. Data will only be transferred to other researchers under a signed data sharing agreement.
  Materials and research data files will be made available, upon request, from the PI. These requests can be made via email (mary.f.brunette@dartmouth.edu).
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing after we complete our analyses, estimated to be in January 2020.
Access Criteria: Investigators wishing to access data will submit a request with an analysis plan, data management plan and data safety plan to the PI. A signed data sharing agreement will be developed prior to release of the data.

REFERENCES:
- [Derived] Brunette MF, Ferron JC, McGurk SR, Williams JM, Harrington A, Devitt T, Xie H. Brief, Web-Based Interventions to Motivate Smokers With Schizophrenia: Randomized Trial. JMIR Ment Health. 2020 Feb 8;7(2):e16524. doi: 10.2196/16524. PMID 32039811

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After participating in an informed consent process, 184 subjects were assessed for eligibility. 11 were ineligible and 11 declined or were unable to proceed with the study for other reasons. 162 were randomized and proceeded to receive an intervention.
Groups:
- Let's Talk About Smoking: These participants were randomized to use the Let's Talk About Smoking website. This web-based intervention (Let's Talk About Smoking) is designed to increase motivation to quit smoking by using evidence-based treatment. Based on the Theory of Planned Behavior [98], the decision support system addresses beliefs that are barriers to cessation and introduces new beliefs that facilitate use of cessation treatment. It uses messages with both gain and loss frames (benefits of use, costs of not using treatment) [140, 141]. It also provides facts with simple text and pictures about risks and benefits for each cessation treatment [142-144], encouraging users to make a choice based on information about treatment options. The system aims to change beliefs and attitudes related to cessation and cessation treatment.
- National Cancer Institute (NCI) Computerized Education: The control intervention that is comparable to previous research - a pamphlet that provides education and advice to quit in computerized form. We have computerized a publicly available educational pamphlet (with advice to quit) for the usual care control condition [162] (Appendix B). This control program is designed with similar usability features to the intervention program, but does not contain any of the features believed to increase the efficacy of our active intervention (interactive assessment and feedback, video role models, etc).
Period: Overall Study
Arm/Group | Let's Talk About Smoking | National Cancer Institute (NCI) Computerized Education
Started | 78 | 84
Completed | 68 | 77
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 4 | 4
Not completed — moved | 1 | 1
Not completed — Lost to Follow-up | 4 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Educational Intervention: Computerized version of the National Cancer Institute (NCI) Educational Pamphlet
  NCI Education
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention | Educational Intervention | Total
Number analyzed (Participants) | 78 | 84 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.62 (11.29) | 44.32 (11.18) | 45.91 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 49 | 59 | 108
Region of Enrollment [Number; unit: participants]
  United States | 78 | 84 | 162
Brief Psychiatric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — A structured assessment of psychopathology severity using structured interview, observation, and record review. Scores may range from 7 to 126.
  units on a scale | 41.79 (11.95) | 40.38 (10.32) | 41.06 (11.11)
Positive and Negative Affect Schedule - Positive [Mean (Standard Deviation); unit: units on a scale] — Self report measure of positive affect. Scores range from 10 (low positive affect) to 50 (high positive affect).
  units on a scale | 22.36 (8.66) | 22.31 (8.48) | 22.33 (8.54)
Positive and Negative Affect Schedule - Negative [Mean (Standard Deviation); unit: units on a scale] — 10 Item self report measure of negative affect. Scores may range from 10 (low negative affect) to 50 (high negative affect).
  units on a scale | 12.04 (9.09) | 12.06 (9.45) | 12.05 (9.25)
Cognition battery Z Scores [Mean (Standard Deviation); unit: units on a scale] — We used a composite score of cognition measures including attention-concentration (Continuous Performance Test), verbal and working memory (Hopkins Verbal Learning Test), and processing speed (Trail Making Test Part A), as well as cognitive flexibility (Trail Making Test Part B) and inhibitory control (Stroop subtest) with measures from the DKEFS (Delis-Kaplan Executive Functioning System).
  For each individual, we normalized each of their scale scores and calculated a mean of these scores. This mean served as the individual's composite cognition score.
  units on a scale | -.029 (0.68) | .016 (0.70) | -.006 (0.69)
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes] — Self-reported number of cigarettes smoked per day.
  cigarettes | 14.48 (9.62) | 14.64 (11.3) | 14.56 (10.49)
Fagerstrom dependence score [Mean (Standard Deviation); unit: units on a scale] — The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. The test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.
  Yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  units on a scale | 5.03 (2.19) | 5.30 (1.80) | 5.16 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Initiated Cessation Treatment
Description: Cessation treatment initiation and engagement will be collected from clinician attendance sheets in the medical record and medical record review for prescriptions. Medication use will be confirmed with self-report of taking medication.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Let's Talk About Smoking | National Cancer Institute (NCI) Computerized Education
Number analyzed (Participants) | 78 | 84
participants | 27 | 36

2. Secondary Outcome: Number of Subjects With Confirmed Abstinence
Description: Biologically confirmed abstinence: we will confirm 7-day point prevalence abstinence at 6 month assessments (self-reported abstinence without any smoking, "not even a puff," for the past 7 days,) with expired carbon monoxide (reading ≤9).
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Let's Talk About Smoking: These participants were randomized to use the Let's Talk About Smoking website. This web-based intervention (Let's Talk About Smoking) is designed to increase motivation to quit smoking by using evidence-based treatment. Based on the Theory of Planned Behavior, the decision support system addresses beliefs that are barriers to cessation and introduces new beliefs that facilitate use of cessation treatment. It uses messages with both gain and loss frames (benefits of use, costs of not using treatment). It also provides facts with simple text and pictures about risks and benefits for each cessation treatment, encouraging users to make a choice based on information about treatment options. The system aims to change beliefs and attitudes related to cessation and cessation treatment.
- National Cancer Institute (NCI) Computerized Education: The control intervention that is comparable to previous research - a pamphlet that provides education and advice to quit in computerized form. We have computerized a publicly available educational pamphlet (with advice to quit), using large font text, limited content per screen, and audio, for the usual care control condition. This control program is designed with similar usability features to the intervention program, but does not contain any of the features believed to increase the efficacy of our active intervention (interactive assessment and feedback, video role models, etc).
Arm/Group | Let's Talk About Smoking | National Cancer Institute (NCI) Computerized Education
Number analyzed (Participants) | 78 | 84
participants | 1 | 6

3. Secondary Outcome: Number of Subjects With a Quit Attempt With 7 or More Days of Self-reported Abstinence
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Intervention | Educational Intervention
Number analyzed (Participants) | 78 | 84
Participants | 13 | 11

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Behavioral Intervention: These participants were randomized to use the Let's Talk About Smoking website. This web-based intervention (Let's Talk About Smoking) is designed to increase motivation to quit smoking by using evidence-based treatment. Based on the Theory of Planned Behavior [98], the decision support system addresses beliefs that are barriers to cessation and introduces new beliefs that facilitate use of cessation treatment. It uses messages with both gain and loss frames (benefits of use, costs of not using treatment) [140, 141]. It also provides facts with simple text and pictures about risks and benefits for each cessation treatment [142-144], encouraging users to make a choice based on information about treatment options. The system aims to change beliefs and attitudes related to cessation and cessation treatment.
- Educational Intervention: The control intervention that is comparable to previous research - a pamphlet that provides education and advice to quit in computerized form. We have computerized a publicly available educational pamphlet (with advice to quit) for the usual care control condition [162] (Appendix B). This control program is designed with similar usability features to the intervention program, but does not contain any of the features believed to increase the efficacy of our active intervention (interactive assessment and feedback, video role models, etc).
Arm/Group | Behavioral Intervention | Educational Intervention
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/84
Other Adverse Events (participants affected / at risk) | 0/78 | 1/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Intervention (N=78) | Educational Intervention (N=84)
Death (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Intervention (N=78) | Educational Intervention (N=84)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes